CLINICAL TRIAL: NCT05235607
Title: Personalized Immune Cell Therapy Targeting Neoantigen of Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PITTN2021
Record Dates: First submitted 2021-12-19; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Carcinoma; Melanoma; Bladder Cancer; Colorectal Cancer
Keywords: Melanoma; Bladder Cancer; Colorectal Cancer; tumor neo-antigen DC vaccine; safety; clinical efficacy
MeSH Terms: conditions — Carcinoma; Melanoma; Urinary Bladder Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor antigen-sensitized vaccine and their sensitized T cells (Experimental): Tumor antigen-sensitized vaccine is administrated, 1- week interval, totally 2 times.
  Then, Neo-antigen DC vaccine and their sensitized T cells are administrated, 2-week interval, totally 5 times.
  Interventions: Biological: Tumor antigen-sensitized DC vaccine and their sensitized T cells subcutaneous administration

INTERVENTIONS:
Biological: Tumor antigen-sensitized DC vaccine and their sensitized T cells subcutaneous administration — subcutaneous administration

SUMMARY:
This single center, single arm and prospective study aimed to establish gene mutation database and select the neoantigens in patients with advanced malignant melanoma, bladder cancer and colorectal cancer. Then, we intended to explore the safety and efficacy of individual tumor antigen-sensitized DC vaccine and their sensitized T cells in these solid cancers.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-75 years
* Pathologically diagnosed advanced (stage IV) malignant melanoma, bladder cancer or colorectal cancer with measurable lesions;
* Failed in the previous standard therapy;
* ECOG PS (Eastern Cooperative Oncology Group performance status) score 0-2 points;
* The estimated survival period is ≥3 months;
* Rehabilitate from previous therapy;
* Adequate organ functions;
* Patient's written informed consent;

Exclusion Criteria:

* Tumor emergencies;
* Abnormal coagulation function;
* Contagious diseases, such as HIV, HBV, HCV infection;
* Mental disorders;
* Concomitant tumors;
* Immunological co-morbidities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as events as assessed by CTCAE v4.0 | 3 months after the last administration of cells
  Number of participants with treatment-related adverse events as events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Number of participants with Overall survival as assessed by RECIST1.1 | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Yan Liu, Principal Investigator — Sichuan University
Locations (1):
- West China Hospital, Chengdu, Sichuan, China